CLINICAL TRIAL: NCT01226901
Title: A Phase I Study of MK-4827 in Patients With Solid Tumor
Brief Title: A Phase I Study of MK-4827 for Treatment of Solid Tumors (MK-4827-005)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Vice President, Late Stage Development Group Leader, Merck Sharp & Dohme Corp
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-4827-005
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Neoplasms; Solid Tumors
Keywords: Poly (ADP-ribose) polymerase (PARP) inhibitor; tumor; cancer
MeSH Terms: conditions — Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-4827 once daily (Experimental): MK-4827
  Interventions: Drug: MK-4827

INTERVENTIONS:
Drug: MK-4827 — MK-4287, 150 mg or 300 mg capsule, orally, once daily in 21 day cycles.

SUMMARY:
This study will evaluate whether oral administration of MK-4827 to participants with advanced solid tumors is generally safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a histologically or cytologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist. There is no limit on the number of prior treatment regimens.
* Participant has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group(ECOG) Performance Scale
* Participant must have adequate organ function (per prespecified laboratory values).

Exclusion Criteria:

* Participant has had major surgery, chemotherapy, radiotherapy, hormonal or biological therapy within 4 weeks (6 weeks for nitrosoureas, mitomycin C, or bevacizumab) prior to entering the study.
* Participant has known central nervous system metastases or a primary central nervous system tumor.
* Participant is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study.
* Participant is known to be Human Immunodeficiency Virus (HIV)-positive.
* Participant with active Hepatitis B or C.
* Participant has symptomatic ascites or pleural effusion.
* Participant has interstitial lung disease as a history or current evidence.
* Participant has known bleeding tendency or coagulation disorder as a history or current evidence, and/or participant is taking any anti-coagulant and/or antiplatelet therapies.
* Participant has uncontrolled persistent or active infection (acute infection which requires antibiotic or anti-fungal treatment).
* Participant has participated in a clinical trial with a known Poly (ADP-ribose) polymerase (PARP) inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) in Cycle 1 | Cycle 1 of treatment (1 cycle = 21 days)
  Dose-limiting toxicities are defined as all adverse experiences that are clearly not related to disease progression or intercurrent illness. In order to be declared a dose-limiting toxicity, an adverse experience must be related (definitely, probably, or possibly) to study therapy.